CLINICAL TRIAL: NCT03548038
Title: Taste Changes With Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Professor, University of Missouri-Columbia
Other Study IDs: 2011543
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-03

CONDITIONS: Taste, Altered
Keywords: taste perception; bariatric surgery; taste preference; weight loss surgery
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Before bariatric surgery, the subject will lightly scrape the inside of their cheek to harvest cells. These cell will be frozen for future DNA extraction and detection of taste receptor genes, T1R2 and T1R3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surgery patients: All subjects will be patients scheduled for bariatric surgery. There is only one arm in this study.
  Interventions: Other: taste test

INTERVENTIONS:
Other: taste test — All subjects will complete a procedure to determine their taste sensitivity to sweet tastants.

SUMMARY:
It is commonly believed that a link exists between BMI and taste perception. One group of researchers observed that women who are obese experience reduced taste sensitivity when compared to normal-weight controls. Others have compared taste sensitivity between lean and obese subjects and found no significant differences. The inconsistencies in these studies demonstrate how much variation in taste sensitivity is possible when different factors are applied in research. Throughout several studies, one element remains constant - bariatric surgery causes appetite aversions. These changes in appetite and food preference likely have a large influence on the overall magnitude of post-surgical weight loss. Although many studies have investigated the changes in taste preference after bariatric surgery, few, if any, have focused on changes in sweet taste perception.

DETAILED DESCRIPTION:
The overall goal of the present project is to determine how future bariatric surgery will affect the taste for sweet liquids. Taste perception will be assessed before surgery (pre-operative, pre-op) and after bariatric surgery, at approximately 1 month. Taste studies will be conducted with solutions prepared freshly before each test using sucrose dissolved in distilled water. Six concentrations of sucrose (table sugar) will be tasted in random order, with the most concentrated solution being roughly the sweetness of soda. The subject is blinded to the concentrations. It is hypothesized that there will be no significant difference in taste perception when pre-op and post-op values are compared. However, the investigators hypothesize that taste preference will identify solutions with lower concentrations post-op.

ELIGIBILITY:
Inclusion Criteria:

* Women who plan to undergo bariatric surgery.
* Age: 21-70y.
* Non-smokers (at least 3 months post smoking cessation).
* Non-diabetic or prediabetic

Exclusion Criteria:

* Subject on a medication known to affect taste perception: Antibiotics, thyroid medications, psychotropic, neurological, and cardiac medications.
* Inability to understand the test instructions.
* Subject has already undergone bariatric surgery

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects will be included.
Study Population: Women aged 21-70 will be recruited from the University of Missouri Bariatric Surgery Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Taste Perception on an Interval Scale | Change from baseline to one month after bariatric surgery
  Taste perception will be assessed by the subjects' responses to varying sucrose solutions. The interval scale begins with "barely detectable" at zero and goes up to "strongest imaginable" at 10. Subjects will be asked to draw an "X" at the location on the graph corresponding to their perception.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Elizabeth Parks, Columbia, Missouri
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bueter M, Miras AD, Chichger H, Fenske W, Ghatei MA, Bloom SR, Unwin RJ, Lutz TA, Spector AC, le Roux CW. Alterations of sucrose preference after Roux-en-Y gastric bypass. Physiol Behav. 2011 Oct 24;104(5):709-21. doi: 10.1016/j.physbeh.2011.07.025. Epub 2011 Jul 30. PMID 21827777
- [Background] Scruggs DM, Buffington C, Cowan GS Jr. Taste Acuity of the Morbidly Obese before and after Gastric Bypass Surgery. Obes Surg. 1994 Feb;4(1):24-28. doi: 10.1381/096089294765558854. PMID 10742759
- [Background] Pepino MY, Finkbeiner S, Beauchamp GK, Mennella JA. Obese women have lower monosodium glutamate taste sensitivity and prefer higher concentrations than do normal-weight women. Obesity (Silver Spring). 2010 May;18(5):959-65. doi: 10.1038/oby.2009.493. Epub 2010 Jan 14. PMID 20075854